CLINICAL TRIAL: NCT06584435
Title: A Single-arm Study of Toripalimab in Adjuvant Therapy After Resection of High-risk Renal Cancer
Brief Title: A Study of Toripalimab in Adjuvant Therapy After Resection of High-risk Renal Cancer
Acronym: TUORA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUORA
Record Dates: First submitted 2024-09-02; First posted 2024-09-04 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-11

CONDITIONS: High-risk Renal Cell Carcinoma
Keywords: High-risk Renal Cell Carcinoma; Toripalimab; Adjuvant therapy
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High risk recurrent renal cell carcinoma patients receiving treatment with Toripalimab (Experimental): Intervention: Toripalimab, a humanized anti-PD-1 monoclonal antibody. Dosage & Administration: Fixed dose of 240 mg via intravenous infusion every 3 weeks (Q3W). Treatment commences within 4-12 weeks post-nephrectomy.
  Treatment Duration: Administered for up to 17 cycles (approximately one year), or until disease recurrence, unacceptable toxicity, or meeting other discontinuation criteria.
  Dose Modification Policy: Dose adjustment is not permitted. Management of specific immune-related adverse events (irAEs) is strictly limited to therapy suspension (with potential resumption after symptom improvement to Grade 0-1) or permanent discontinuation, as per protocol-specified guidelines.
  Key Assessments: Includes regular tumor imaging (CT/MRI) every 12 weeks, comprehensive safety monitoring, and quality of life evaluations.
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — Drug Profile: Toripalimab , a humanized IgG4 anti-PD-1 monoclonal antibody with unique structural features.
  Key Differentiators:
  Dosing Protocol: Fixed 240mg Q3W regimen (not weight-based) Administration: 30-minute IV infusion with mandatory 0.2μm filtration Dose Policy: Strictly no dose adjustment permitted - only suspension/discontinuation allowed for toxicity management
  Unique Features:
  Binding Specificity: Toripalimab targets a unique conformational epitope on the PD-1 receptor's CC' loop, differentiated from pembrolizumab (binding FG loop) and nivolumab (binding BC loop). This results in varied steric hindrance effects and potentially distinct immune activation kinetics.The specific binding interface may influence receptor internalization dynamics and duration of pathway blockade, contributing to toripalimab's characteristic clinical activity and safety profile observed in prior studies.

SUMMARY:
The goal of this clinical trial is to learn if the drug toripalimab (an anti-PD-1 antibody) works to prevent cancer recurrence in patients with high-risk renal cell carcinoma after they have had surgery to remove the kidney (nephrectomy). The study will also learn about the safety of toripalimab in this setting.The main questions the study aims to answer are:

1. Does treatment with toripalimab after nephrectomy increase the time patients live without their cancer returning (disease-free survival) compared to what would be expected without this treatment?
2. What medical problems (side effects) do participants have when receiving toripalimab? This is a single-arm study, meaning all participants in the trial will receive the study drug, toripalimab.. Researchers will monitor participants over time to see if the outcomes with toripalizumab are better than what is historically known for similar patients who only had surgery.

Participants in this study will:

1. Receive toripalimab by intravenous (IV) infusion once every 3 weeks for up to about one year ( 17 doses).
2. Visit the clinic regularly for check-ups, which will include:

Imaging scans (like CT or MRI) of the chest, abdomen, and pelvis every 12 weeks to check for cancer recurrence.

Blood and urine tests to monitor safety. Questionnaires about their quality of life and symptoms. Be followed for a long period after treatment ends to track overall survival and long-term health.

DETAILED DESCRIPTION:
1. Study Background and Rationale Renal cell carcinoma (RCC) carries a substantial risk of recurrence post-nephrectomy, particularly in patients with intermediate-high risk, high risk, or M1 no evidence of disease (NED) status following metastasectomy. The phase III KEYNOTE-564 clinical trial demonstrated that adjuvant therapy with pembrolizumab, an anti-PD-1 antibody, significantly improved disease-free survival (DFS) compared to placebo in this patient population, establishing a new therapeutic standard. Building upon this landmark finding, the present study aims to investigate the efficacy and safety of toripalimab, another anti-PD-1 monoclonal antibody, within a similar clinical context. This single-arm, phase II trial seeks to evaluate whether toripalimab can provide comparable clinical benefits, including reduced recurrence risk and improved survival outcomes, for patients with high-risk RCC following complete surgical resection, while thoroughly assessing its safety profile.
2. Study Objectives

   Primary Objectives:

   To evaluate the efficacy of adjuvant toripalimab as measured by investigator-assessed Disease-Free Survival (DFS) and Overall Survival (OS).

   Secondary Objectives:

   To assess the safety and tolerability profile of adjuvant toripalimab and patient-reported outcomes (PROs) using quality of life questionnaires..
3. Trial Design and Methodology This is a single-center, prospective, single-arm, Phase II clinical trial. The design leverages the positive signal observed in the KEYNOTE-564 trial to explore the potential of a similar immunotherapeutic agent, toripalimab, in a real-world setting at a major academic center. The study will enroll patients who have undergone nephrectomy and are within the 4 to 12-week postoperative window. Treatment involves intravenous administration of toripalimab at a fixed dose of 240 mg every three weeks, for a planned treatment duration of approximately one year (17 cycles), mirroring the treatment schedule found effective in the precedent trial. Treatment will continue until disease recurrence, unacceptable toxicity, or other protocol-defined discontinuation criteria are met. The single-arm design is chosen to efficiently characterize the activity and safety of toripalimab in this specific adjuvant setting, with outcomes referenced against historical controls and the results of prior pivotal studies.
4. Study Procedures and Assessments

   The assessment schedule is structured to closely monitor for efficacy and safety signals, consistent with the standards set by recent practice-changing trials. Key procedures include:

   Screening Period (Within 4 weeks prior to treatment initiation):
   * Informed consent process.
   * Confirmation of diagnosis and high-risk status via central pathology review .
   * Tumor imaging via CT or MRI of the chest, abdomen, and pelvis to confirm no evidence of disease post-surgery.
   * Collection of archival tumor tissue from nephrectomy/metastasectomy.
   * Physical examination, vital signs, ECOG performance status assessment.
   * Clinical laboratory tests: hematology, serum chemistry, thyroid function, coagulation profile, urinalysis.
   * Viral serology testing (HBV, HCV, HIV).
   * Pregnancy test for women of childbearing potential (WOCBP).
   * Baseline quality of life assessments (EORTC QLQ-C30 and FKSI-15).

   Treatment Period (Each cycle is 3 weeks):
   * Pre-dose assessments (Day 1 of each cycle): Vital signs, directed physical exam, assessment of adverse events (AEs) and concomitant medications.
   * Toripalimab administration: IV infusion on Day 1 of each cycle.
   * Laboratory tests: Hematology and serum chemistry at every cycle; urinalysis and thyroid function tests periodically as specified in the protocol.
   * Tumor imaging: CT/MRI scans of chest, abdomen, and pelvis will be performed every 12 weeks (± 7 days) from the date of treatment to assess for disease recurrence.
   * Quality of Life (QoL) assessments: EORTC QLQ-C30 and FKSI-15 questionnaires will be administered at predefined cycles and at the end of treatment.

   Post-Treatment Follow-up Period:
   * Safety Follow-up Visit: Occurs 30 days (± 7 days) after the last dose of toripalimab for ongoing AE monitoring.
   * Efficacy Follow-up: After treatment discontinuation (without disease recurrence), patients will continue tumor imaging assessments every 12 weeks (Year 1-3), then every 24 weeks (Years 4+) until disease recurrence, start of new anticancer therapy, or study end.
   * Survival Follow-up: Overall survival status will be assessed via telephone or clinic visit every 12 weeks (± 7 days) until death, withdrawal of consent, or the end of the study.
5. Endpoints The endpoints are selected to align with the established efficacy parameters in adjuvant RCC immunotherapy trials, facilitating a meaningful evaluation of toripalimab's benefit-risk profile.

   Primary Endpoint:
   * Disease-Free Survival (DFS) , defined as the time from randomization to the first documented local or distant recurrence or death from any cause.
   * Overall Survival (OS): Defined as the time from randomization to death from any cause.

   Secondary Endpoints: Include incidence and severity of adverse events (AEs/SAEs) graded by CTCAE v5.0, and changes from baseline in PRO scores.
6. Statistical Considerations The sample size is planned to be 40-100 participants. The analysis will be primarily descriptive for this single-arm study. Efficacy analyses (DFS, OS) will be performed on the Full Analysis Set (FAS) using Kaplan-Meier methodology. Safety analyses will be conducted on the Safety Set (SS). The results will be contextualized with reference to existing data from the adjuvant RCC treatment landscape, including findings from the KEYNOTE-564 trial.

ELIGIBILITY:
1. INCLUSION CRITERIA

   Participants must meet ALL of the following criteria to be eligible for study enrollment:

   1.1 Informed Consent Capable of giving signed informed consent； Willing to comply with all study procedures； Signed and dated written informed consent obtained prior to any study-specific procedures.

   1.2 Age and Sex Age ≥18 years at time of consent； Male and female participants eligible. 1.3 Disease Characteristics Histologically confirmed renal cell carcinoma with clear cell component; Must have undergone nephrectomy with complete resection; No evidence of residual tumor confirmed by imaging;

   Must meet at least ONE of the following high-risk criteria:

   pT2,with Fuhrman Grade IV or sarcomatoid,N0,M0;pT3/4,N0M0 (any grade);Any T classification with N1,M0;Post nephrectomy(total/partial) plus complete resection of metastasis, M1 NED.

   1.4 Brain Metastasis No suspected or confirmed active brain metastases. 1.5 Performance Status Eastern Cooperative Oncology Group (ECOG) performance status 0-1. 1.6 Organ Function (within 14 days prior to enrollment, without transfusion or growth factor support)

   Hematopoietic function:

   Absolute neutrophil count ≥1,500/mm³; Platelet count ≥100,000/mm³; Hemoglobin ≥9.0 g/dL (5.6 mmol/L)

   Hepatic function:

   Total bilirubin ≤1.5 × ULN; AST and ALT ≤1.5 × ULN

   Renal function:

   Serum creatinine ≤1.5 mg/dL; OR creatinine clearance ≥60 mL/min (Cockcroft-Gault formula) 1.7 Contraception Females of childbearing potential must use medically approved contraception during treatment and for 3 months after last dose; Negative serum or urine pregnancy test within 7 days prior to randomization for women of childbearing potential; Non-lactating females; Males with female partners of childbearing potential must use effective contraception during treatment and for 3 months after last dose 1.8 Compliance Voluntarily agrees to participate by signing informed consent; Willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
2. EXCLUSION CRITERIA

   Participants meeting ANY of the following criteria will be excluded from study participation:

   2.1 Prior Therapy Previous radiotherapy, chemotherapy, targeted therapy, long-term or high-dose hormone therapy, or any immune checkpoint inhibitor treatment.

   2.2 Concurrent Malignancy History of or current concurrent malignancy (except adequately treated basal cell carcinoma of skin, carcinoma in situ of cervix, etc.).

   2.3 Allergy and Prior Immunotherapy Previous treatment with other PD-1/PD-L1 inhibitors; Known hypersensitivity to macromolecular protein preparations or any PD-1 inhibitor components.

   2.4 Autoimmune Disease Active autoimmune disease or history of autoimmune disease; Exceptions:Controlled type 1 diabetes, hypothyroidism requiring only hormone replacement, skin diseases not requiring systemic treatment (vitiligo, psoriasis), or childhood asthma in complete remission without intervention in adulthood.

   2.5 Immunosuppressive Therapy Current use of immunosuppressants (e.g., systemic corticosteroids >10 mg/day prednisone equivalent) for immunosuppressive purposes, continued within 2 weeks prior to enrollment.

   2.6 Cardiovascular Disease

   Poorly controlled cardiac clinical symptoms or diseases, including:

   NYHA Class II or higher heart failure; Unstable angina pectoris; Myocardial infarction within 1 year; Clinically significant arrhythmias requiring treatment 2.7 Coagulation Function Abnormal coagulation function with bleeding tendency; Current thrombolytic or anticoagulant therapy; 2.8 Gastrointestinal Disease

   Current active gastrointestinal diseases including:

   Esophageal varices; Active ulcers; Inflammatory bowel disease; Risk of perforation or bleeding; 2.9 Hemorrhage and Thrombosis Events History of or current severe hemorrhage, hemoptysis, or thrombotic events within 12 months.

   2.10 Infection Active infection requiring systemic therapy; Unexplained fever >38.5°C during screening or before first dose; Congenital or acquired immunodeficiency, including HIV infection or active hepatitis 2.11 Other Medical Conditions History of severe pulmonary fibrosis, interstitial pneumonia, radiation pneumonia; Live vaccination within 4 weeks prior to study treatment; History of psychotropic drug abuse, alcoholism, or drug addiction 2.12 Administrative Reasons Participation in another clinical study or within 1 month after completion of previous clinical study; Any condition that, in the investigator's judgment, may lead to early study termination affecting participant safety or data quality
3. WITHDRAWAL CRITERIA

Participants will be withdrawn from study treatment if ANY of the following occurs:

3.1 Participant Request Participant or legal representative requests withdrawal 3.2 Disease Progression Confirmed disease progression 3.3 Intolerable Toxicity Occurrence of intolerable toxicities 3.4 Investigator Judgment Investigator determines continued participation may harm the participant 3.5 Protocol Violations Pregnancy Loss to follow-up Major protocol violation 3.6 Treatment Delay Any cause leading to treatment delay >2 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) as Assessed by Investigator | From enrollment until the first documented disease recurrence, distant metastasis, or death from any cause (whichever occurs first), assessed up to 60 months
  Disease-Free Survival is defined as the time from enrollment to the first documented occurrence of any of the following events:
  Local recurrence of renal cell carcinoma (confirmed by imaging) Distant metastasis of renal cell carcinoma (confirmed by imaging) Death from any cause Participants without documented DFS events at the time of analysis will be censored at the date of their last tumor assessment. Tumor assessments will be performed using computed tomography (CT) or magnetic resonance imaging (MRI) according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 guidelines.

SECONDARY OUTCOMES:
Overall Survival (OS) | From enrollment until death from any cause, assessed up to 120 months
  Overall Survival is defined as the time from enrollment to death from any cause. Participants who are alive at the time of analysis will be censored at the last known alive date. Survival status will be collected through regular follow-up contacts every 12 weeks (± 7 days) until death, withdrawal of consent, or the end of the study, whichever occurs first.
Incidence and Severity of Adverse Events | At the following predefined visit time points: first dose (baseline), each subsequent cycle treatment day, and the 90-day safety follow-up visit after the last dose.
  Safety and tolerability will be assessed through:
  * Incidence, severity, and relationship to study treatment of all adverse events (AEs)
  * Serious adverse events (SAEs) and adverse events leading to treatment discontinuation
  * Laboratory abnormalities (hematology, clinical chemistry, urinalysis)
  * Vital signs measurements and physical examination findings
  * Electrocardiogram (ECG) parameters
  * All AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0. Immune-related adverse events (irAEs) will be specifically monitored and managed according to protocol-specified guidelines.
Health-Related Quality of Life Assessment | Baseline, every 12 weeks during treatment (up to 17 cycles), at treatment discontinuation, and every 12 weeks during follow-up until disease recurrence (up to 60 months).
  Quality of life will be evaluated using validated patient-reported outcome (PRO) instruments:
  EORTC QLQ-C30: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 items FKSI-DRS: Functional Assessment of Cancer Therapy-Kidney Symptom Index-Disease-Related Symptoms The EORTC QLQ-C30 assesses global health status and quality of life across multiple domains including physical, role, emotional, cognitive, and social functioning. The FKSI-DRS specifically measures disease-related symptoms in renal cell carcinoma patients. Changes from baseline in scale scores will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Changyi Changyi, MD,PhD, Principal Investigator — Tianjin Medical University Second Hospital
Locations (1):
- Changyi Quan, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
1. Data Scope De-identified individual participant data (IPD) Clinical study report protocols
  2. Data Specifications Clinical Datasets: Demographic/ efficacy (response, survival)/ safety (adverse events) data Documentation: Informed consent templates and complete study protocols Standards: CDISC SDTM/ADaM formatted datasets
  3. Access Process Timeline: Available within 18 months after trial completion Platform: Access via designated data sharing portal Review: Scientific review committee approval required
  4. Usage Terms Purpose: Academic non-commercial research use only Requirements: Signed data sharing agreements mandatory Restrictions: No commercial use or re-identification attempts
  5. Technical Details Format: Analysis-ready datasets with metadata Support: Provided documentation and limited technical support
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Availability Start Date: Individual participant data and supporting documents will become available for sharing 24 months after the primary results publication of the main trial outcomes.
  Data Availability Period: The data will remain accessible for a period of 5 years from the initial sharing date. During this timeframe, qualified researchers may submit requests and access the data through the designated platform.
  Extension Policy: After the initial 5-year period, the availability of the data will be re-evaluated annually. Data may remain accessible beyond this period based on continued scientific interest, resource availability, and platform sustainability.
  Data Updates: The shared datasets represent the final, locked database from the completed clinical trial. No additional updates or amendments to the core dataset are anticipated. However, corrected versions may be released if critical errors are identified, with clear version control maintained.
Access Criteria: 1. Eligible Data Requestors Academic researchers from accredited institutions Regulatory and government health authorities Pharmaceutical company researchers (for non-commercial research) Other qualified scientific researchers with legitimate research inquiries
  2. Accessible Data and Documents De-identified individual participant data Study protocol and statistical analysis plan Annotated case report forms Clinical study report (sanitized) Data dictionaries and metadata documentation
  3. Data Access Process 3.1 Application Requirements Submission of research proposal through designated portal Detailed statistical analysis plan required Proof of institutional review board approval Signed data sharing agreement 3.2 Review and Approval Independent review by scientific committee 60-day standard review period Evaluation based on scientific merit and feasibility Approval notification with access credentials
  4. Permitted Research Uses Conducting meta-analyses

REFERENCES:
- [Result] Chen J, Ji T, Zhao J, Li G, Zhang J, Jin R, Liu J, Liu X, Liang X, Huang D, Xie A, Lin H, Cang Y, Cai X. Sorafenib-resistant hepatocellular carcinoma stratified by phosphorylated ERK activates PD-1 immune checkpoint. Oncotarget. 2016 Jul 5;7(27):41274-41284. doi: 10.18632/oncotarget.8978. PMID 27129180
- [Result] Fukuda T, Kamai T, Masuda A, Nukui A, Abe H, Arai K, Yoshida K. Higher preoperative serum levels of PD-L1 and B7-H4 are associated with invasive and metastatic potential and predictable for poor response to VEGF-targeted therapy and unfavorable prognosis of renal cell carcinoma. Cancer Med. 2016 Aug;5(8):1810-20. doi: 10.1002/cam4.754. Epub 2016 Jun 12. PMID 27292320
- [Result] Chen Y, Ramjiawan RR, Reiberger T, Ng MR, Hato T, Huang Y, Ochiai H, Kitahara S, Unan EC, Reddy TP, Fan C, Huang P, Bardeesy N, Zhu AX, Jain RK, Duda DG. CXCR4 inhibition in tumor microenvironment facilitates anti-programmed death receptor-1 immunotherapy in sorafenib-treated hepatocellular carcinoma in mice. Hepatology. 2015 May;61(5):1591-602. doi: 10.1002/hep.27665. Epub 2015 Mar 20. PMID 25529917
- [Result] Choueiri TK, Figueroa DJ, Fay AP, Signoretti S, Liu Y, Gagnon R, Deen K, Carpenter C, Benson P, Ho TH, Pandite L, de Souza P, Powles T, Motzer RJ. Correlation of PD-L1 tumor expression and treatment outcomes in patients with renal cell carcinoma receiving sunitinib or pazopanib: results from COMPARZ, a randomized controlled trial. Clin Cancer Res. 2015 Mar 1;21(5):1071-7. doi: 10.1158/1078-0432.CCR-14-1993. Epub 2014 Dec 23. PMID 25538263
- [Result] Hughes PE, Caenepeel S, Wu LC. Targeted Therapy and Checkpoint Immunotherapy Combinations for the Treatment of Cancer. Trends Immunol. 2016 Jul;37(7):462-476. doi: 10.1016/j.it.2016.04.010. Epub 2016 May 20. PMID 27216414
- [Result] Voron T, Colussi O, Marcheteau E, Pernot S, Nizard M, Pointet AL, Latreche S, Bergaya S, Benhamouda N, Tanchot C, Stockmann C, Combe P, Berger A, Zinzindohoue F, Yagita H, Tartour E, Taieb J, Terme M. VEGF-A modulates expression of inhibitory checkpoints on CD8+ T cells in tumors. J Exp Med. 2015 Feb 9;212(2):139-48. doi: 10.1084/jem.20140559. Epub 2015 Jan 19. PMID 25601652
- [Result] Hato T, Zhu AX, Duda DG. Rationally combining anti-VEGF therapy with checkpoint inhibitors in hepatocellular carcinoma. Immunotherapy. 2016;8(3):299-313. doi: 10.2217/imt.15.126. Epub 2016 Feb 11. PMID 26865127
- [Result] Abdel-Wahab N, Shah M, Suarez-Almazor ME. Adverse Events Associated with Immune Checkpoint Blockade in Patients with Cancer: A Systematic Review of Case Reports. PLoS One. 2016 Jul 29;11(7):e0160221. doi: 10.1371/journal.pone.0160221. eCollection 2016. PMID 27472273
- [Result] Boutros C, Tarhini A, Routier E, Lambotte O, Ladurie FL, Carbonnel F, Izzeddine H, Marabelle A, Champiat S, Berdelou A, Lanoy E, Texier M, Libenciuc C, Eggermont AM, Soria JC, Mateus C, Robert C. Safety profiles of anti-CTLA-4 and anti-PD-1 antibodies alone and in combination. Nat Rev Clin Oncol. 2016 Aug;13(8):473-86. doi: 10.1038/nrclinonc.2016.58. Epub 2016 May 4. PMID 27141885
- [Result] Wu C, Zhu Y, Jiang J, Zhao J, Zhang XG, Xu N. Immunohistochemical localization of programmed death-1 ligand-1 (PD-L1) in gastric carcinoma and its clinical significance. Acta Histochem. 2006;108(1):19-24. doi: 10.1016/j.acthis.2006.01.003. Epub 2006 Mar 13. PMID 16530813
- [Result] Gao Q, Wang XY, Qiu SJ, Yamato I, Sho M, Nakajima Y, Zhou J, Li BZ, Shi YH, Xiao YS, Xu Y, Fan J. Overexpression of PD-L1 significantly associates with tumor aggressiveness and postoperative recurrence in human hepatocellular carcinoma. Clin Cancer Res. 2009 Feb 1;15(3):971-9. doi: 10.1158/1078-0432.CCR-08-1608. PMID 19188168
- [Result] Mu CY, Huang JA, Chen Y, Chen C, Zhang XG. High expression of PD-L1 in lung cancer may contribute to poor prognosis and tumor cells immune escape through suppressing tumor infiltrating dendritic cells maturation. Med Oncol. 2011 Sep;28(3):682-8. doi: 10.1007/s12032-010-9515-2. Epub 2010 Apr 6. PMID 20373055
- [Result] Robert C, Ribas A, Wolchok JD, Hodi FS, Hamid O, Kefford R, Weber JS, Joshua AM, Hwu WJ, Gangadhar TC, Patnaik A, Dronca R, Zarour H, Joseph RW, Boasberg P, Chmielowski B, Mateus C, Postow MA, Gergich K, Elassaiss-Schaap J, Li XN, Iannone R, Ebbinghaus SW, Kang SP, Daud A. Anti-programmed-death-receptor-1 treatment with pembrolizumab in ipilimumab-refractory advanced melanoma: a randomised dose-comparison cohort of a phase 1 trial. Lancet. 2014 Sep 20;384(9948):1109-17. doi: 10.1016/S0140-6736(14)60958-2. Epub 2014 Jul 15. PMID 25034862
- [Result] Davies M. New modalities of cancer treatment for NSCLC: focus on immunotherapy. Cancer Manag Res. 2014 Feb 3;6:63-75. doi: 10.2147/CMAR.S57550. eCollection 2014. PMID 24520205
- [Result] Hamid O, Carvajal RD. Anti-programmed death-1 and anti-programmed death-ligand 1 antibodies in cancer therapy. Expert Opin Biol Ther. 2013 Jun;13(6):847-61. doi: 10.1517/14712598.2013.770836. Epub 2013 Feb 19. PMID 23421934
- [Result] Wolchok JD, Hoos A, O'Day S, Weber JS, Hamid O, Lebbe C, Maio M, Binder M, Bohnsack O, Nichol G, Humphrey R, Hodi FS. Guidelines for the evaluation of immune therapy activity in solid tumors: immune-related response criteria. Clin Cancer Res. 2009 Dec 1;15(23):7412-20. doi: 10.1158/1078-0432.CCR-09-1624. Epub 2009 Nov 24. PMID 19934295
- [Result] Zielinski C, Knapp S, Mascaux C, Hirsch F. Rationale for targeting the immune system through checkpoint molecule blockade in the treatment of non-small-cell lung cancer. Ann Oncol. 2013 May;24(5):1170-9. doi: 10.1093/annonc/mds647. Epub 2013 Feb 7. PMID 23393121
- [Result] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Result] Hamid O, Robert C, Daud A, Hodi FS, Hwu WJ, Kefford R, Wolchok JD, Hersey P, Joseph RW, Weber JS, Dronca R, Gangadhar TC, Patnaik A, Zarour H, Joshua AM, Gergich K, Elassaiss-Schaap J, Algazi A, Mateus C, Boasberg P, Tumeh PC, Chmielowski B, Ebbinghaus SW, Li XN, Kang SP, Ribas A. Safety and tumor responses with lambrolizumab (anti-PD-1) in melanoma. N Engl J Med. 2013 Jul 11;369(2):134-44. doi: 10.1056/NEJMoa1305133. Epub 2013 Jun 2. PMID 23724846
- [Result] McDermott DF, Atkins MB. PD-1 as a potential target in cancer therapy. Cancer Med. 2013 Oct;2(5):662-73. doi: 10.1002/cam4.106. Epub 2013 Jul 21. PMID 24403232
- [Result] Brahmer JR, Drake CG, Wollner I, Powderly JD, Picus J, Sharfman WH, Stankevich E, Pons A, Salay TM, McMiller TL, Gilson MM, Wang C, Selby M, Taube JM, Anders R, Chen L, Korman AJ, Pardoll DM, Lowy I, Topalian SL. Phase I study of single-agent anti-programmed death-1 (MDX-1106) in refractory solid tumors: safety, clinical activity, pharmacodynamics, and immunologic correlates. J Clin Oncol. 2010 Jul 1;28(19):3167-75. doi: 10.1200/JCO.2009.26.7609. Epub 2010 Jun 1. PMID 20516446
- [Result] Blank C, Mackensen A. Contribution of the PD-L1/PD-1 pathway to T-cell exhaustion: an update on implications for chronic infections and tumor evasion. Cancer Immunol Immunother. 2007 May;56(5):739-45. doi: 10.1007/s00262-006-0272-1. Epub 2006 Dec 29. PMID 17195077
- [Result] Qu HX, Zhao LP, Zhan SH, Geng CX, Xu L, Xin YN, Jiang XJ. Clinicopathological and prognostic significance of programmed cell death ligand 1 (PD-L1) expression in patients with esophageal squamous cell carcinoma: a meta-analysis. J Thorac Dis. 2016 Nov;8(11):3197-3204. doi: 10.21037/jtd.2016.11.01. PMID 28066599
- [Result] Hara H, Tahara M, Daiko H, Kato K, Igaki H, Kadowaki S, Tanaka Y, Hamamoto Y, Matsushita H, Nagase M, Hosoya Y. Phase II feasibility study of preoperative chemotherapy with docetaxel, cisplatin, and fluorouracil for esophageal squamous cell carcinoma. Cancer Sci. 2013 Nov;104(11):1455-60. doi: 10.1111/cas.12274. Epub 2013 Oct 18. PMID 23991649
- [Result] von Dobeln GA, Klevebro F, Jacobsen AB, Johannessen HO, Nielsen NH, Johnsen G, Hatlevoll I, Glenjen NI, Friesland S, Lundell L, Yu J, Nilsson M. Neoadjuvant chemotherapy versus neoadjuvant chemoradiotherapy for cancer of the esophagus or gastroesophageal junction: long-term results of a randomized clinical trial. Dis Esophagus. 2019 Feb 1;32(2). doi: 10.1093/dote/doy078. PMID 30137281
- [Result] Stahl M, Walz MK, Riera-Knorrenschild J, Stuschke M, Sandermann A, Bitzer M, Wilke H, Budach W. Preoperative chemotherapy versus chemoradiotherapy in locally advanced adenocarcinomas of the oesophagogastric junction (POET): Long-term results of a controlled randomised trial. Eur J Cancer. 2017 Aug;81:183-190. doi: 10.1016/j.ejca.2017.04.027. PMID 28628843
- [Result] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Result] Yang H, Liu H, Chen Y, Zhu C, Fang W, Yu Z, Mao W, Xiang J, Han Y, Chen Z, Yang H, Wang J, Pang Q, Zheng X, Yang H, Li T, Lordick F, D'Journo XB, Cerfolio RJ, Korst RJ, Novoa NM, Swanson SJ, Brunelli A, Ismail M, Fernando HC, Zhang X, Li Q, Wang G, Chen B, Mao T, Kong M, Guo X, Lin T, Liu M, Fu J; AME Thoracic Surgery Collaborative Group. Neoadjuvant Chemoradiotherapy Followed by Surgery Versus Surgery Alone for Locally Advanced Squamous Cell Carcinoma of the Esophagus (NEOCRTEC5010): A Phase III Multicenter, Randomized, Open-Label Clinical Trial. J Clin Oncol. 2018 Sep 20;36(27):2796-2803. doi: 10.1200/JCO.2018.79.1483. Epub 2018 Aug 8. PMID 30089078
- [Result] Bhansali MS, Vaidya JS, Bhatt RG, Patil PK, Badwe RA, Desai PB. Chemotherapy for carcinoma of the esophagus: a comparison of evidence from meta-analyses of randomized trials and of historical control studies. Ann Oncol. 1996 Apr;7(4):355-9. doi: 10.1093/oxfordjournals.annonc.a010601. PMID 8805926

DOCUMENTS (3):
  • Study Protocol (2022-10-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT06584435/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT06584435/SAP_001.pdf
  • Informed Consent Form (2022-10-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT06584435/ICF_002.pdf